CLINICAL TRIAL: NCT02177851
Title: The Optimization of Bioavailability From Iron Supplements: Examinations of Different Supplementation Regimens Including Hepcidin Profiles
Brief Title: The Optimization of Bioavailability From Iron Supplements: Study 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: FeSupp_Hep-2
Record Dates: First submitted 2014-06-25; First posted 2014-06-30 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2015-09

CONDITIONS: Iron Deficiency; Anemia; Iron Deficiency Anemia
Keywords: Iron bio-availability; Hepcidin; Iron absorption
MeSH Terms: conditions — Iron Deficiencies; Anemia; Anemia, Iron-Deficiency

ARMS (2):
- Single oral iron supplement per day (120 mg) (Experimental): Single oral iron dose of 120 mg per day for 3 consecutive days
  Interventions: Dietary Supplement: Single oral iron dose of 120 mg per day for 3 consecutive days
- B.i.d. oral iron supplement (2x 60 mg) (Active Comparator): Two oral iron doses of 60 mg per day (morning + afternoon) for 3 consecutive days
  Interventions: Dietary Supplement: Two oral iron doses of 60 mg per day (morning + afternoon) for 3 consecutive days

INTERVENTIONS:
Dietary Supplement: Single oral iron dose of 120 mg per day for 3 consecutive days
  Arms: Single oral iron supplement per day (120 mg)
Dietary Supplement: Two oral iron doses of 60 mg per day (morning + afternoon) for 3 consecutive days
  Arms: B.i.d. oral iron supplement (2x 60 mg)

SUMMARY:
Iron deficiency (ID) with or without anaemia (IDA) is a major public health problem worldwide, especially in women of reproductive age and young children. Iron supplementation is an effective strategy to prevent and treat ID and IDA. There is a lack of data on iron bioavailability from different supplementation regimens and how to optimize bioavailability in a cost-effective and patient-friendly way. The daily supplementation with 1-4 mg Fe/kg body weight for 3 months is reported to be the most effective method to rapidly increase iron stores in subjects with ID and IDA. In IDA patients, medical practitioners often prescribe supplementation regimens with 120 mg iron per day split into 2 doses with 60 mg iron, arguing that the splitting would increase iron bioavailability compared with one single high dose. However, there is no scientific evidence for this assumption; to the contrary, results from a recent study suggest that iron bioavailability from a second supplementation dose of iron after a first supplementation dose of iron is impaired due to increased hepcidin levels. To address this bioavailability issue, the present study will determine iron absorption from 120 mg iron administered for 3 consecutive days and compare it with that from 2 doses of 60 mg iron per day administered for 3 consecutive days. The investigators hypothesize that the iron bioavailability from the single daily dose will be lower than that from the 2 doses. By measuring also hepcidin, this study will provide important insights on the iron bioavailability from a single dose of iron and on the same amount iron split into two doses (b.i.d. administration).

ELIGIBILITY:
Inclusion Criteria:

* Female, 18 to 45 years old,
* Serum Ferritin levels <20 µg/L,
* Normal body Mass Index (18.5-25 kg/m2),
* Body weight <65 kg,
* Signed informed consent

Exclusion Criteria:

* Anaemia (Hb < 11.7 g/dL),
* Elevated c-reactive protein or alpha1 glycoprotein concentrations >5.0 mg/L, >1.0 g/L, respectively,
* Any metabolic, gastrointestinal kidney or chronic disease such as diabetes, renal failure, hepatic dysfunction, hepatitis, hypertension, cancer or cardiovascular diseases (according to the participants own statement),
* Continuous/long-term use of medication during the whole studies (except for contraceptives),
* Consumption of mineral and vitamin supplements within 2 weeks prior to 1st supplement administration,
* Blood transfusion, blood donation or significant blood loss (accident, surgery) over the past 4 months,
* Earlier participation in a study using stable iron isotopes,
* Known hypersensitivity or allergy to iron supplements,
* Women who are pregnant or breast feeding,
* Intention to become pregnant during the course of the studies,
* Lack of safe contraception, defined as: Female participants of childbearing potential, not using and not willing to continue using a medically reliable method of contraception for the entire study duration, such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices, or who are not using any other method considered sufficiently reliable by the investigator in individual cases.
* Known or suspected non-compliance, drug or alcohol abuse,
* Inability to follow the procedures of the studies, e.g. due to language problems, psychological disorders, dementia, etc. of the participant,
* Participation in another study with investigational drug within the 30 days preceding and during the present studies,
* Enrolment of the investigator, his/her family members, employees and other dependent persons

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-06; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Iron bio-availability (%) from oral iron supplementation (3x 120 mg) | 3 days
  Iron bioavailability will be assessed with stable isotopic labels. The shift in the isotopic ratio in human whole blood will be measured with Inductively coupled plasma mass spectrometry (ICP-MS).
Serum hepcidin concentrations on the 1st day of iron supplementation | 1 day
Iron bio-availability (%) from oral iron supplementation (6x 60 mg) | 6 days
  Iron bioavailability will be assessed with stable isotopic labels. The shift in the isotopic ratio in human whole blood will be measured with Inductively coupled plasma mass spectrometry (ICP-MS).
Serum hepcidin concentrations on the 2nd day of iron supplementation | 2 days
Serum hepcidin concentrations on the 3rd day of iron supplementation | 3 days
Serum hepcidin concentrations on the 4th day of iron supplementation | 4 days
Serum hepcidin concentrations on the 5th day of iron supplementation | 5 days
Serum hepcidin concentrations on the 6th day of iron supplementation | 6 days

CONTACTS AND LOCATIONS:
Locations (1):
- Human Nutrition Laboratory, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Stoffel NU, Cercamondi CI, Brittenham G, Zeder C, Geurts-Moespot AJ, Swinkels DW, Moretti D, Zimmermann MB. Iron absorption from oral iron supplements given on consecutive versus alternate days and as single morning doses versus twice-daily split dosing in iron-depleted women: two open-label, randomised controlled trials. Lancet Haematol. 2017 Nov;4(11):e524-e533. doi: 10.1016/S2352-3026(17)30182-5. Epub 2017 Oct 9. PMID 29032957